CLINICAL TRIAL: NCT03854812
Title: Magnesium Sulphate Versus Fentanyl as Adjuvants to Propofol for Monitored Anesthesia Care During Burr-hole Surgery for Chronic Subdural Hematoma: Randomized Clinical Trial
Brief Title: Magnesium Sulphate Versus Fentanyl Sedation During Burr-hole Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Lecturer of Anesthesia, surgical intensive care and pain mangement, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N28-2018
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Monitored Anesthesia Care
Keywords: magnesium sulphate; fentanyl; propofol; monitored anesthesia care; burr-hole evacuation; chronic subdural hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Magnesium Sulfate; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): magnesium sulphate as adjuvant to propofol
  Interventions: Drug: Magnesium Sulphate; Drug: Propofol
- Group F (Active Comparator): fentanyl as adjuvant to propofol
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Magnesium Sulphate — a loading of 50 mg/kg in 15 minutes of Magnesium sulphate, and will be followed by continuous infusion at 1 ml/kg/h of 15 mg/ml solution
  Other Names: magnesium sulfate
  Arms: Group M
Drug: Fentanyl — loading of 1 mcg/kg in over 15 minutes of fentanyl then will receive continuous infusion starting at 1 ml /kg/h. of 0.5 mcg/ml solution
  Arms: Group F
Drug: Propofol — 0.5-1.5 mg/kg bolus of propofol over 10 minutes to achieve target Ramsay sedation scale (RSS) of 3 (respond to command), if RSS afterwards does not reach 3 a supplementary bolus dose of 0.2 mg/kg propofol will be given to the patients, and will be followed by 1-2.5 mg/kg/hr infusion to maintain Intraoperative BIS readings between 60 - 80

SUMMARY:
MgSO4 was found to reduce the perioperative anesthetic and analgesic requirements when used as an adjuvant to general anesthesia. Fentanyl is a potent opioid and used as adjuvant to other sedatives in awake craniotomy procedure. No study, to the best of our knowledge had evaluated fentanyl continuous infusion, nor MgSo4 infusion as adjuvant sedative agents to propofol during Burr-hole surgery. The aim of this study is to evaluate and compare MgSO4 versus fentanyl continuous infusions for conscious sedation in patients undergoing burr hole surgery for evacuation of subdural hematoma with local infiltration.

DETAILED DESCRIPTION:
All participants or their proxy will be informed about the anesthetic techniques and the operative procedure and will provide written informed consent before enrollment in the study.

The eligible patients will be randomly divided by computer designed lists and then will be concealed in closed envelopes into the two study groups. A research assistant who will not be involved in patient management will be responsible for opening the envelope, group assignment and drugs preparation.

Anesthetic management Pre-induction No premedication will be administered. Upon arrival to the operating theater, an intravenous (IV) cannula will be placed, and standard monitors, including 5-lead electrocardiogram, noninvasive arterial blood pressure monitor, and pulse oximetry, will be applied. Oxygen supplementation at fraction of inspired oxygen (FiO2) of 0.35 will be achieved through a suitable air entrainment mask. Bispectral index (BIS: apparatus info) will be applied before starting the drug infusions and will be used for maintenance of sedation during operation.

Induction of anesthesia Group M (n=17): will receive a loading of 50 mg/kg in 15 minutes of Magnesium sulphate, and will be followed by continuous infusion at 1 ml/kg/h of 15 mg/ml solution Group F (n=17): will receive a loading of 1 mcg/kg in over 15 minutes of fentanyl then will receive continuous infusion starting at 1 ml /kg/h. of 0.5 mcg/ml solution Both groups will be given 0.5-1.5 mg/kg bolus of propofol over 10 minutes to achieve target Ramsay sedation scale (RSS) of 3 (respond to command), if RSS afterwards does not reach 3 a supplementary bolus dose of 0.2 mg/kg propofol will be given to the patients, and will be followed by 1-2.5 mg/kg/hr infusion to maintain Intraoperative BIS readings between 60 - 80.

Intraoperative management After achieving the target sedation level (RSS of 3), surgeons will infiltrate the surgical site with 20 mL of a local anesthetic solution containing 10 mL of 0.5% bupivacaine and 10 mL of 2% lidocaine with adrenaline at least 5 minutes before surgical incision. After performing burr-hole craniotomy soaked pledgets with lidocaine will be applied to anaesthetize the dura, the dura will be then opened, and the hematoma will be evacuated. The Infusion of sedatives will be ceased after skin closure.

Intraoperative patient's movements (defined as those which may interfere with the surgical conduct such as twisting of hand and/or leg and head mobility) will be managed by reassurance and support for 30 seconds. However, when movements continue, a bolus dose of propofol of 0.5 mg/kg will be given then infusion dose will be increased till the maximum dose (2.5mg/kg/hr) to regain BIS sedation score between 60-80. If the patient starts to move again the same sequence will be repeated. Minute movements of other body parts as well as movements of fingers or toes that unlikely to hinder the operative intervention, will be deemed insignificant to be documented.

Induction of general anesthesia will be only indicated if satisfactory surgical conditions will not be attained by the rescue propofol.

Intraoperative bradycardia and tachycardia (defined as heart rate (HR) < 45 bpm or > 120 bpm respectively) will be treated with intravenous atropine 0.2 mg, or propranolol 0.5-1 mg respectively. Hypertension and hypotension (defined as a more than 25% increase or decrease from baseline respectively) will be treated with nitroglycerine (0.1-10 mcg/min) or ephedrine (5 mg) respectively.

Postoperative management All patients will be transferred to the post-anesthesia care unit (PACU) after surgery where they will be closely monitored with the aid of five-lead electrocardiography and non-invasive arterial blood pressure, peripheral oxygen saturation (SpO2), and respiratory rate readings using an automated system for 24 h after surgery. Postoperative pain intensity will be assessed using VAS score at 1, 2, 3 and 6 hours after PACU admission. If VAS score exceeds 3, 30 mg of ketorolac will be administered.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral, chronic subdural hematoma,
* aged above 50 years,
* american society of anesthesiologist-physical status (ASA-PS) grade I-II,
* Glasgow coma scale of 14-15.

Exclusion Criteria:

* Patients with hypertension (Systolic blood pressure > 160 mmHg),
* bradycardia (<50 bpm),
* ischemic heart disease,
* second- or third-degree heart block,
* long-term abuse of or addiction to opioids, and sedative-hypnotic drugs (>6 months),
* allergy to study drugs
* neuropsychiatric diseases
* patients with predicted difficult airway
* patients with history of obstructive sleep apnea
* patients with deviation in the surgical technique
* inadequacy of local anesthesia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
average systolic blood pressure | after induction of conscious sedation till end of procedure
  mmgh

SECONDARY OUTCOMES:
ephedrine use | after induction of conscious sedation till end of procedure
  mg
Total amount of Propofol consumption | after induction of conscious sedation till end of procedure
  mg
Total number of intraoperative patient's movements | after induction of conscious sedation till end of procedure
  defined as those likely to interfere with surgical procedure such as bending of hand and/or leg and movement of head
Systolic blood pressure | upon arrival at the operating room, after induction of conscious sedation, at skin incision, at 1,2,5,10,15 min and 10 min after skin incision, every 15 minutes intraoperative, on arrival at PACU, 5,10,15,30 min and 1 hour at the PACU
  mmgh
Diastolic blood pressure | upon arrival at the operating room, after induction of conscious sedation, at skin incision, at 1,2,5,10,15 min and 10 min after skin incision, every 15 minutes intraoperative, on arrival at PACU, 5,10,15,30 min and 1 hour at the PACU
  mmgh
Heart rate | upon arrival at the operating room, after induction of conscious sedation, at skin incision, at 1,2,5,10,15 min and 10 min after skin incision, every 15 minutes intraoperative, on arrival at PACU, 5,10,15,30 min and 1 hour at the PACU
  bpm
Surgeon satisfaction score | 30 minutes after the end of the surgery
  1, extremely dissatisfied; 2, not satisfied but able to manage; 3, satisfied; 4, extremely satisfied.
Ramsay sedation scale | 15 and 30 minutes postoperative
  Ramsey 1 Anxious, agitated, restless Ramsey 2 Cooperative, oriented, tranquil Ramsey 3 Responsive to commands only If Asleep Ramsey 4 Brisk response to light glabellar tap or loud auditory stimulus Ramsey 5 Sluggish response to light glabellar tap or loud auditory stimulus Ramsey 6 No response to light glabellar tap or loud auditory stimulus
Visual Analogue Scale (VAS) for pain | at 15 minutes, 30 minutes, 1hr, 2 hrs. 3hrs and 6 hrs after PACU admission
  10 cm horizontal line on which the patient's pain intensity is represented by a point between the extremes of 0=no pain at all and 10 cm = worst pain imaginable."
atropine use | after induction of conscious sedation till end of procedure
  mg
first rescue analgesic during 1 hour post operative | 1 hour postoperative
  incidence of patients requiring analgesics
postoperative nausea and vomiting | first 24 hours in the postoperative period
  incidence

CONTACTS AND LOCATIONS:
Overall Officials: Maha mostafa, MD, Principal Investigator — kasr el aini
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rodriguez-Rubio L, Nava E, Del Pozo JSG, Jordan J. Influence of the perioperative administration of magnesium sulfate on the total dose of anesthetics during general anesthesia. A systematic review and meta-analysis. J Clin Anesth. 2017 Jun;39:129-138. doi: 10.1016/j.jclinane.2017.03.038. Epub 2017 Apr 7. PMID 28494889
- [Background] Sinha PK, Koshy T, Gayatri P, Smitha V, Abraham M, Rathod RC. Anesthesia for awake craniotomy: a retrospective study. Neurol India. 2007 Oct-Dec;55(4):376-81. doi: 10.4103/0028-3886.33308. PMID 18040111
- [Background] Gignac E, Manninen PH, Gelb AW. Comparison of fentanyl, sufentanil and alfentanil during awake craniotomy for epilepsy. Can J Anaesth. 1993 May;40(5 Pt 1):421-4. doi: 10.1007/BF03009510. PMID 8513521